Study Title: A Multi-centred, Randomised, Open Label, Placebo-controlled, Two-period Crossover Study to Evaluate 4-hour Esophageal pH Change in GERD Patients After Administration of Compound Sodium Alginate Double Action Tablets or Placebo Tablets

ClinicalTrials.gov ID: NCT01872897

Final Statistical Analysis Plan, dated 25-Feb-2014

Changes to Planned Statistical Analyses Form, dated 19-Mar-2014

Changes to Planned Statistical Analyses Form, dated 08-May-2014

Changes to Planned Statistical Analyses Form, dated 17-Jul-2014



# STATISTICAL ANALYSIS PLAN

# **GA1202**

A MULTI-CENTRED, RANDOMISED, OPEN LABEL, PLACEBO-CONTROLLED, TWO-PERIOD CROSSOVER STUDY TO EVALUATE 4-HOUR ESOPHAGEAL PH CHANGE IN GERD PATIENTS AFTER ADMINISTRATION OF COMPOUND SODIUM ALGINATE **DOUBLE ACTION CHEWABLE TABLETS OR MATCHING PLACEBO TABLETS** 

**AUTHOR:** 

VERSION NUMBER AND DATE: V5.1(FINAL), 25FEB2014

Document:

Reckitt Benckiser GA1202 Statistical Analysis Plan

Author:

Version Number: Version Date:

[25Feb2014] Reference: CS WI BS005

Final 5.1

Template No: CS TP BS016 - Revision 3


Effective Date: 01May2012





# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan Final V5.1 (Date 25Feb2014) for Protocol <<GA1202 >> Dated 01Mar2013

| | | Name | Signature | is appropriate |
|---------|-----------|------------------------|-----------|----------------|
| Author: | | | | |
| | Position: | Manager, Biostatistics | | |
| ř | Company: | Quintiles | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

Approved By:

Position: Statistical Manager

Company: Reckitt Benckiser Brands Limited

Document:

Reckitt Benckiser GA1202 Statistical Analysis Plan

Author:

Version Number: Version Date: Final 5.1 [25Feb2014]

Template No: CS\_TP\_BS016 - Revision 3

Reference: CS\_WI\_BS005

Effective Date: 01May2012






# **MODIFICATION HISTORY**

| Unique<br>Identifier<br>for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| 0.1 | 16Apr2013 | | Not Applicable – First Version |
| 0.2 | 30Jul2013 | | Update per internal comments |
| 0.3 | 16Aug2013 | | Update per internal comments |
| 0.4 | 19Aug2013 | | Update per internal comments |
| 0.5 | 20Aug2013 | | Update per internal comments |
| 1.0 | 20Aug2013 | | Update to draft version 1.0 and sent to sponsor for review |
| 1.1 | 02SEP2013 | | Update per sponsor's comment |
| 1.2 | 06Sep2013 | | Update per internal review comment |
| 2.0 | 06Sep2013 | | Update to draft version 2.0 and sent to sponsor for review |
| 3.0 | 210ct2013 | | Update per sponsor's comment |
| 3.1 | 23Oct2013 | | Update per sponsor's comment |
| 4.0 | 25Oct2013 | | Update to final version 4.0 |
| 5.0 | 10Jan2014 | | Update to present the concomitant medication by ATC level. |
| 5.1 | 25Feb2014 | Update FAS definition Change listings (16.2.3.1-16.2.3.8) to be presented on FAS instead of all patients. Updated list of tables and listings per sponsor's comments. | |

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan

Effective Date: 01May2012

Author: Version Number: Final 5.1
Version Date: [25Feb2014]

Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






# **LIST OF ABBREVIATIONS AND DEFINITION OF TERMS**

| AE | Adverse event |
|--------|----------------------------------------------|
| ANOVA | Analysis of Variance |
| ATC | Anatomical Therapeutic Chemical |
| BLQ | Below the lower limit of quantification |
| CI | Confidence Interval |
| CRF | Case report form |
| FAS | Full analysis set |
| GERD | Gastro-esophageal reflux disease |
| IMP | Investigational medicinal product |
| ITT | Intention-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NIMP | Non-investigational medicinal product |
| PP | Per protocol |
| PT | Preferred term |
| SAE | Serious adverse event |
| SOC | System organ class |
| SAP | Statistical analysis plan |
| SI | International System |
| ULQ | Upper limit of quantification |
| WHO | World Health Organization |

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan

Effective Date: 01May2012

Author: Version Number: Version Date:

Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005


Final 5.1

[25Feb2014]





# **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 8 |
|------|--------------------------------------------------------|----|
| 2. | STUDY OBJECTIVES | 8 |
| 2.1. | Primary Objective | 8 |
| 2.2. | Secondary Objectives | 8 |
| 3. | STUDY DESIGN | 9 |
| 3.1. | General Description | 9 |
| 3.2. | Schedule of Events | 9 |
| 4. | FINAL ANALYSIS | 9 |
| 5. | ANALYSIS SETS | 9 |
| 5.1. | Full Analysis Set [FAS] | 9 |
| 5.2. | Safety Population | 10 |
| 5.3. | Intent-to-treat [ITT] Population | 10 |
| 5.4. | Per Protocol [PP] Population | 10 |
| 6. | GENERAL CONSIDERATIONS | 10 |
| 6.1. | Reference Start Date and Study Day | 10 |
| 6.2. | Baseline | 11 |
| 6.3. | Retests, Unscheduled Visits and Early Termination Data | 11 |
| 6.4. | Statistical Tests | 11 |
| 6.5. | Common Calculations | 11 |
| 6.6. | Software Version | 12 |

Document:

Reckitt Benckiser GA1202 Statistical Analysis Plan

Author:

Version Number: Version Date: Final 5.1 [25Feb2014]

Template No: CS\_TP\_BS016 - Revision 3

Effective Date: 01May2012

Reference: CS\_WI\_BS005 





| 7. | STATISTICAL CONSIDERATIONS | | 12 |
|---|---|---|---|
| 7.1 | Adjustments for Covariates and Factors to be Include | ed in Analyses | 12 |
| 7.1. | Multicenter Studies | | 12 |
| 7.2. | Missing data | | 12 |
| 7.3. | Examination of Subgroups | | 12 |
| 7.4. | Multiple Comparisons/ Multiplicity | | 13 |
| 8. | OUTPUT PRESENTATIONS | | 13 |
| 9. | DISPOSITION AND WITHDRAWALS | | 13 |
| 10. | DEMOGRAPHIC AND OTHER BASELINE ( | CHARACTERISTICS | 13 |
| 10.1. | Derivations | | 14 |
| 11. | MEDICAL HISTORY | | 14 |
| 12. | CONCOMITANT ILLNESSES | | 14 |
| 13. | PRIOR AND CONCOMITANT MEDICATIO | N AND THERAPIES | 15 |
| 14. | STUDY MEDICATION EXPOSURE & COMI | PLIANCE | 15 |
| 14.1. | Derivations | | 16 |
| <b>15</b> . | EFFICACY OUTCOMES | | 16 |
| 15.1. | Primary Efficacy | | 16 |
| 15.1 | • | | |
| 15.1 | , , | | |
| 15.1 | | | |
| 15.1 | 1.4 Sensitivity Analysis of Primary Efficacy Variable | | 17 |
| 15.2. | Secondary Efficacy | | 17 |
| 15.2 | 2.1 Secondary Efficacy Variables | | 17 |
| 15.2 | <u> </u> | | 18 |
| Docum | - | | |
| Author | | Version Number: | Final 5.1 |

Template No: CS\_TP\_BS016 - Revision 3

Effective Date: 01May2012

Reference: CS\_WI\_BS005 





| 15.2 | 2.3 Analyses of Secondary Efficacy Variables | 19 |
|---|---|---|
| 15.2 | 2.4 Sensitivity Analyses of Secondary Efficacy Variables | 19 |
| 16 | SAFETY OUTCOMES | 19 |
| 16.2 | Adverse Events | 19 |
| 16.2 | 2.1 Adverse Events | 20 |
| 1 | 6.2.1.1 Severity | 21 |
| 1 | 6.2.1.2 Relationship to Study Medication | 21 |
| 16.2 | 2.2 Adverse Events leading to Dose Change or Discontinuation of Study Medication | 21 |
| 16.2 | 2.3 Serious Adverse Events | 21 |
| 16.2 | 2.4 Adverse Events Leading to Death | 21 |
| 16.3 | Death | 21 |
| 16.4 | Laboratory Evaluations | 22 |
| 16.5 | ECG Evaluations | 22 |
| 16.6 | Vital Signs | 23 |
| 16.7 | Physical Examination | 23 |
| 16.8 | References | 23 |
| 17 | LIST OF TABLES | 23 |
| 18 | LIST OF LISTINGS | 25 |
| APPI | ENDIX 1 LIST OF LABORATORY ASSESSMENTS | 26 |

Reckitt Benckiser GA1202 Statistical Analysis Plan Document:

Author: Version Number: Final 5.1 Version Date: [25Feb2014]

Reference: CS\_WI\_BS005 Template No: CS\_TP\_BS016 - Revision 3

 Effective Date: 01May2012



### 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for Protocol GA1202. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 2, amendment 1, dated 4Jul2013.

# 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVE

The primary objective is to compare the time during the 4 hour post dosing period where the pH is below pH 4 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets.

# 2.2. SECONDARY OBJECTIVES

The following secondary endpoints will also be evaluated:

- Percentage of time during the 4 hour post dosing period with pH below pH 5
- Number of occasions during the 4 hour post dosing period when pH falls below pH 4
- Number of occasions during the 4 hour post dosing period when pH falls below pH 5
- Number of reflux episodes during the 4 hour post dosing period with pH below pH 4 for at least 5 minutes
- Percentage of time during the first hour post dosing with pH below pH 4
- Percentage of time during the first hour post dosing with pH below pH 5
- Number of occasions during the first hour post dosing when pH falls below pH 4
- Number of occasions during the first hour post dosing when pH falls below pH 5
- The longest reflux time during the 4 hour post dosing period (i.e. the longest period with pH below pH 4)
- The DeMeester scores during the 4 hour post dosing period.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan

Effective Date: 01May2012

Author: Version Number: Final 5.1 Version Date: [25Feb2014]

Template No: CS TP BS016 - Revision 3 Reference: CS WI BS005




# 3. STUDY DESIGN

## 3.1. GENERAL DESCRIPTION

This is a multi-centre, randomised, open-label, placebo-controlled, two-period crossover study. Forty - four (44) patients are planned to be enrolled in this study to ensure that thirty six (36) patients complete it. After signing a written informed consent, patients will undergo a screening period up to 10 days. Patients who satisfy the study entry requirements within 10 days of consent, will be randomised to receive either four Compound Sodium Alginate Double Action Chewable Tablets or four matching placebo tablets following placement of a pH electrode and a standardised refluxogenic meal.

Upon completion of the 4-hour post-dose pH monitoring period patients will be instructed to begin taking supplied Compound Sodium Alginate Double Action Chewable Tablets (two tablets four times daily) for 7 days. Patients will return after the 7 day period for repeat catheter insertion and pH monitoring, receiving the alternative randomised treatment.

# 3.2. SCHEDULE OF EVENTS

Schedule of assessments can be found in Section 3.10 of the protocol.

# 4. FINAL ANALYSIS

All final, planned analyses identified in this SAP will be performed by Quintiles Biostatistics following Reckitt Benckiser's Authorization of this SAP, Database Lock and Sponsor Authorization of Analysis Sets.

# 5. ANALYSIS SETS

Agreement and authorization of patients included/excluded from each analysis set will be conducted at data review meeting before database lock.

# 5.1. FULL ANALYSIS SET [FAS]

All patients enrolled (e.g. those assigned randomization number) in the study will be included in full analysis set (FAS).

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005

Effective Date: 01May2012





# **5.2.** SAFETY POPULATION

All patients who are subjected to any invasive procedures and/or take at least one dose of study medication will be included in safety population.

# 5.3. INTENT-TO-TREAT [ITT] POPULATION

All patients who take at least one dose of study medication and have evaluable pH monitoring data for at least 1 hour post-dosing will be included into intent-to-treat (ITT) population.

# 5.4. PER PROTOCOL [PP] POPULATION

The inclusion/exclusion from per protocol (PP) population will be confirmed during data review meeting, but will include patients who satisfied following criteria and did not experience any major protocol violations in ITT population: patients who adhered to the inclusive/exclusive criteria; did not take any prohibited medication which would interfere with evaluation of drugs in the study period; attended visits within the specified visit windows and had complete pH monitoring data for 4 hour post-dosing for both pH monitoring visits.

A major violation of the protocol is defined as any violation of the protocol that is considered to affect the efficacy results and may include the following:

- When a randomization error or administration of the wrong study medication occurred;
- When the patient did not satisfy the inclusion/exclusion criteria;
- When the patient had taken prohibited concomitant medications;
- When the patient failed to attend visit at specified visit windows;
- When the efficacy (4 hour post-dosing monitoring) evaluation was not completed for either monitoring visits.

Protocol violations will be categorized before database lock and will be summarized (by treatment sequence group and overall) and listed.

## 6. GENERAL CONSIDERATIONS

## 6.1. Reference Start Date and Study Day

Study Day will be calculated from the reference start date, and will be used to show start/stop day of assessments and events.

Reference start date (Day 0) is defined as the day of first dose of study medication.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005

Effective Date: 01May2012 





Study Day = (date of event – reference start date).

In the situation where the event date is partial or missing, Study Day, and any corresponding durations will appear partial or missing in the listings.

Randomization date will be considered as the same date of randomization visit, that is, visit 2.

# 6.2. BASELINE

Unless otherwise specified, baseline value refers to the tests or measurements recorded at Visit 1, screening visit. If a particular test or measurement was repeated after Visit 1, screening visit, then the baseline value is defined as the last non-missing measurement taken prior to Visit 2, Day 0 (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered pre-baseline, but Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline.

For patients randomized but not treated, baseline is defined as the last non-missing measurement taken on or before the baseline visit date.

# 6.3. RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

In general, for by-visit summaries, data recorded at the nominal visit will be presented. Unscheduled measurements will not be included in by-visit summaries. In the case of a retest (same visit number assigned), the latest available measurement for that visit will be used for by-visit summaries.

Early termination data will be mapped to the next available visit number for by-visit summaries.

Listings will include scheduled, unscheduled, retest and early discontinuation data.

# **6.4. STATISTICAL TESTS**

The default significant level will be (5%); confidence intervals (CIs) will be 95% and all tests will be two-sided, unless otherwise specified in the description of the analyses.

# 6.5. COMMON CALCULATIONS

For quantitative measurements, change from baseline will be calculated as:

• Test Value at Visit X – Baseline Value

Effective Date: 01May2012

Log transformed (natural logarithm) of efficacy data (or another transformation) might be used in the statistical models if after inspection of the data it is considered necessary. This decision will be undertaken in collaboration with the sponsor.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






# 6.6. SOFTWARE VERSION

All analyses will be conducted using SAS version 9.2 or higher.

# 7. STATISTICAL CONSIDERATIONS

# 7.1 ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The following factors are used in the analyses. For details of their inclusion in the models, see section 15.1.3.

- Treatment (Study medication and matching placebo tablets)
- Dose visit (Visit 2 and Visit 3)
- Subject
- Treatment sequence (Group A: Patients take study medication at Visit 2 and matching placebo tablets and Visit 3. Group B: Patients take study medication at Visit 3 and matching placebo tablets at Visit 2.

### 7.1. MULTICENTER STUDIES

This study will be conducted at two or more hospital sites. The 4-hour pH endpoints will be summarized separately for each center. Center will not be included as a factor in any of the statistical models because the study has a cross-over design

## 7.2. MISSING DATA

Effective Date: 01May2012

Patients who withdraw from the study will not be replaced.

Unless otherwise specified, all analysis will be based on the number of non-missing observations, i.e. patients with missing information will not be included in the denominator when calculating percentages. If relevant for categorical tabulations, missing values will be treated as another category, so that all tabulations involving this variable will also include a row or column as appropriate to indicate the number of patients for whom the variable was recorded as a missing value.

For AEs, partial or missing dates and times will not be imputed, and this will be listed as originally reported in the Case Report Form (CRF).

## 7.3. EXAMINATION OF SUBGROUPS

No subgroup analyses will be performed for this study.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






# 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

Since there is only one primary analysis, no multiple comparison adjustments will be used.

# 8. OUTPUT PRESENTATIONS

The table and listing templates provided with this SAP describe the conventions for presentation of data in outputs, and presentations for this study and therefore the format and content of the summary tables, figures and listings to be provided by Quintiles Biostatistics.

## 9. DISPOSITION AND WITHDRAWALS

The number of patients who provided informed consent, as well as those who were eligible at Visit 1 and Visit 2 (met all inclusion criteria and not met all exclusion criteria) will be summarized overall. The number of patients who completed the study, the number of patients who withdrew prematurely from the study, the reasons for withdrawals and the number of patients in the FAS, Safety, ITT and PP population (see Section 4 for population definitions) will be summarized for each treatment sequence group and overall. Listings on patient completion/withdrawal information, as well as eligibility details will be reported

Major protocol violations will be summarized by treatment sequence group and overall. Furthermore the number of patients to be excluded from each population together with reasons of exclusion will be summarized. Details on major protocol violations as well as population classification information will be listed.

## 10. Demographic and other Baseline Characteristics

Demographic data and other baseline characteristics will be summarized by treatment sequence group and overall for all patients in FAS.

No statistical testing will be carried out for demographic or other baseline characteristics.

The following demographic and other baseline characteristics will be reported for this study:

- Age (years) calculated relative to date of consent
- Race
- Sex
- Height
- Weight

Counts and percentages will be displayed for patients with smoking habits (no, yes, former), alcohol/drug use (no, yes) and drugs of abuse history; summary statistics (mean, median, minimum, maximum and standard deviation) will be provided for the continuous variables including height, weight, age, smoking/drinking years and amount. These data will also be listed.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005

Effective Date: 01May2012 





including the severity and frequency of heartburn. In addition, 12 lead ECG and a standard hospital endoscopy examination will be conducted at baseline as part of the screening procedures. The following Information on ECG and endoscopy will be presented by summary statistics:

Summary statistics will be presented for patients' baseline Gastro-esophageal reflux disease (GERD) symptoms,

ECG:

Whether ECG is performed

Interpretation of ECG results

**Endoscopy:** 

Whether endoscopy performed

Whether local anaesthetic throat spray administered

Whether a sedative administered

Any abnormalities presented in endoscopy

If the patient has erosive GERD

If the patient have hiatus hernia and diameter of the hernia

Other baseline characteristics such as laboratory evaluations, vital signs, and physical examination are specified in section 16.3, 16.5 and 16.6 respectively.

# 10.1. DERIVATIONS

Effective Date: 01May2012

Age = Date of Informed Consent - Date of Birth (rounded down to the nearest whole year)

#### 11. MEDICAL HISTORY

Medical History conditions are defined as those conditions which stopped prior to or at screening visit. Medical history information will be coded using version 16.0 of Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary and presented for all patients in FAS by system organ class (SOC) and preferred term (PT), for each treatment sequence group and overall.

#### **12. CONCOMITANT ILLNESSES**

Concomitant illnesses are conditions other than GERD which are ongoing before or on the day of last dose of Investigational Medicinal Product (IMP), or stopped after screening visit but before or on the day of last dose of IMP. Concomitant Illnesses will be captured from Medical History and Current Status form in CRF, and will be coded using MedDRA version 16.0 and presented for all patients in safety population by SOC and PT, for each treatment sequence group and overall.

Reckitt Benckiser GA1202 Statistical Analysis Plan Document:

Author: Version Number: Final 5.1 Version Date: [25Feb2014]

Template No: CS TP BS016 - Revision 3 Reference: CS WI BS005






# 13. PRIOR AND CONCOMITANT MEDICATION AND THERAPIES

Medications will be coded using World Health Organization (WHO) Drug Dictionary Enhanced version dated 01Mar2013 and tabulated using the Anatomical Therapeutic Chemical (ATC) classification system, under Level 3 and Level 4 for the FAS (for prior and concomitant medications separately)

- 'Prior' medications are medications which started and stopped prior to first dose of study medication.
- 'Concomitant' medications are medications which:
  - o started prior to, on or after first dose of study medication
  - o AND ended on or after first dose of study medication or were ongoing at the end of the study.

# 14. STUDY MEDICATION EXPOSURE & COMPLIANCE

At each of the pH monitoring visits, patients will be administered four Compound Sodium Alginate Double Action Chewable Tablets or four matching placebo tablets under the supervision of the Investigator or his or her delegate. No measurement on medication compliance will be performed.

In addition, all patients will then receive Compound Sodium Alginate Double Action Chewable Tablets (two tablets four times daily) as Non-investigational Medicinal Product (NIMP) for symptomatic treatment. The number of tablets dispensed and returned will be recorded in CRF and presented by table and listing.

The following information regarding whether the patients fulfill each requirement prior to pH monitoring and the time interval from each procedure to taking treatment will be summarized by treatment sequence group:

Requirement prior to pH monitoring:

Not taken symptomatic treatment for GERD (antacids etc) in the 24 hours prior to pH monitoring

Abstain from alcohol 24 hours prior to the test meal

Fast for a minimum of 4 hours prior to insertion of manometry probe

Insert manometry probe to aid positioning of esophageal pH sensor prior to consuming test meal

Consume the entire reflux provoking meal

Record pH from 30 minutes prior to dosing to 4 hours post dosing

Time interval from each procedure to taking treatment:

Position pH electrode (90 mins before treatment)

Eat test meal (60 mins before treatment)

Activate pH monitoring data logger and Record (30 mins before treatment)

Stop pH monitoring (4 hour post dose)

Effective Date: 01May2012

The calculation of time interval is provided in section 14.1

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005




# 14.1. DERIVATIONS

Time interval from each procedure to taking treatment (minutes) is calculated by

Time of the procedure – Time when patient takes treatment

#### **15**. **EFFICACY OUTCOMES**

# 15.1. PRIMARY EFFICACY

#### 15.1.1. PRIMARY EFFICACY VARIABLE

The primary efficacy endpoint is the percentage of time during the 4 hour post dosing period with pH below pH 4 for Compound Sodium Alginate Double Action Chewable Tablets versus matching placebo tablets. This variable is collected on the "Results of 4-hour pH Monitoring" page in CRF.

### 15.1.2. Missing Data Methods for Primary Efficacy Variable

If less than 2 hours post-dosing monitoring result for this variable is available, for whatever reason, the derived variable will be considered missing. If 2 or more hours post-dosing monitoring data is available, the parameter will be derived by multiplying by the factor (4 hours / time with data available). Any data recorded more than 4 hours post-dosing will be ignored when deriving these parameter.

The table below shows the implementation of adjustment rules under different monitoring duration scenarios.

| Monitoring Duration(End of pH monitoring – taking treatment) | Percentage of time with pH<4 during the monitoring period (data directly from database) | Number of hours<br>with pH<4 during<br>the monitoring<br>period | Adjustment factor | Adjusted percentage with pH<4 over 4 hours |
|---|---|---|---|---|
| 240 mins (4 hours) | 80.0% | 240 mins | 1 | 80.0% |
| 230 mins (<4 hours) | 80.0% | 230*80% mins | 240/230 | 230*80%*240/23<br>0/240=80.0% |
| 90 mins (<2 hours) | 20.0% | 90*20% mins | NA | missing |

# 15.1.3 PRIMARY ANALYSIS OF PRIMARY EFFICACY VARIABLE

The primary endpoint will be analysed primarily using a linear mixed model with treatment, dosing visit and

Reckitt Benckiser GA1202 Statistical Analysis Plan Document:

Author: Version Number: Final 5.1 Version Date: [25Feb2014]

Template No: CS TP BS016 - Revision 3 Reference: CS WI BS005


Effective Date: 01May2012





treatment sequence as fixed effects and patient nested within treatment sequence as a random effect. The primary analysis is to test the null hypothesis that there is no difference between treatment, Least square means (with 95% CI) corresponding to the two treatments will be presented. Descriptive statistics will also be presented for the primary endpoint by treatment for each dosing visit and overall. The effects for dosing visit and treatment sequence will also be assessed.

The following SAS core code will be used.

```
proc mixed data=XXX method=REML;
  class treatment visit sequence subID;
  model Y= treatment visit sequence /ddfm=kenwardroger;
  random subID(sequence);
  lsmeans treatment/diff cl;
run;
```

SAS output from Mixed procedure will be sent to the sponsor to assist with the model assumptions review.

The linear mixed model for the primary endpoint is based on the assumption that the percentage of time with pH<4 within each treatment sequence group is normally distributed. To test this assumption, a qualitative residual analysis will be performed. If there is a major departure from the assumptions of normality or heteroscedasticity of residuals, then further analysis using transformed data might be performed if deemed necessary. If the analysis based on the transformed data still rises reasonable concerns about validity of the tests then the Wilcoxon Rank-Sum test will be used to compare the dosing visit difference (dosing visit 1 – dosing visit 2) between treatment sequence groups to represent the treatment comparison.

The primary efficacy analysis will be performed for the ITT population using adjusted 4-hour data based on the imputation rule specified in section 15.1.2.

#### 15.1.4 Sensitivity Analysis of Primary Efficacy Variable

A sensitivity analysis will be conducted on the primary endpoint using the PP population.

If the percentage of missing data for the primary endpoint is greater than 10% (data from > 10% patients is not recorded exactly at 4 hours (+/- 5 minutes), an additional complete case sensitivity analysis will be conducted, using only the observed 4-hour (+/- 5 minutes) data.

## 15.2. SECONDARY EFFICACY

### 15.2.1 SECONDARY EFFICACY VARIABLES

The secondary endpoints are:

Effective Date: 01May2012

Percentage of time during the 4 hour post dosing period with pH below pH 5

Number of occasions during the 4 hour post dosing period when pH falls below pH 4

Number of occasions during the 4 hour post dosing period when pH falls below pH 5

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






Number of reflux episodes during the 4 hour post dosing period with pH below pH 4 for at least 5 minutes

Percentage of time during the first hour post dosing with pH below pH 4

Percentage of time during the first hour post dosing with pH below pH 5

Number of occasions during the first hour post dosing when pH falls below pH 4

Number of occasions during the first hour post dosing when pH falls below pH 5

The longest reflux time during the 4 hour post dosing period (i.e. the longest period with pH below pH 4)

The DeMeester scores during the 4 hour post dosing period.

The secondary efficacy analyses will be performed for the ITT population.

#### 15.2.2 Missing Data Methods for Secondary Efficacy Variables

Missing data for the percentage of time during the 4 hour post dosing period with pH below pH 5 due to early termination of recording will be derived in the same way as for the primary efficacy variable.

For the following secondary efficacy variables:

- Number of occasions during the 4 hour post dosing period when pH falls below pH 4
- Number of occasions during the 4 hour post dosing period when pH falls below pH 5
- Number of reflux episodes during the 4 hour post dosing period with pH below pH 4 for at least 5minutes

If less than 2 hours post-dosing monitoring result for these variables is available, for whatever reason, the derived variable will be considered missing. If 2 or more hours post-dosing pH data is available then the variable will be multiplied by 4 / (hours of post-dosing pH data available). Any data recorded more than 4 hours post-dosing will be ignored when deriving these parameters.

The table below shows the implementation of adjustment rules (take number of occasions as an example) under different monitoring duration scenarios.

| Monitoring Duration(End of pH monitoring – taking treatment) | Number of occasions with pH<4 during the monitoring period (data directly from database) | Adjustment factor | Adjusted occasion with pH<4 over 4 hours |
|---|---|---|---|
| 240 mins (4 hours) | 2 | 1 | 2 |
| 230 mins (<4 hours) | 2 | 240/230 | 2*240/230=2.09 |
| 90 mins (<2 hours) | 1 | NA | missing |

Missing data for other secondary endpoints due to early termination of recording will not be derived.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005

Effective Date: 01May2012





Reckitt Benckiser

#### 15.2.3 Analyses of Secondary Efficacy Variables

The analysis methods for all secondary endpoints will be identically to those described for the primary endpoint in 15.1.3.

#### 15.2.4 Sensitivity Analyses of Secondary Efficacy Variables

Sensitivity analyses will be conducted on the secondary endpoints using the PP population.

If the percentage of missing data for the secondary variables listed in section 15.2.2 is greater than 10% (data from > 10% patients is not recorded exactly at 4 hours +/- 5 minutes), an additional complete case sensitivity analysis will be conducted, using only the observed 4-hour (+/- 5 minutes) data.

# **16** SAFETY OUTCOMES

All outputs for safety outcomes will be based on the Safety Population.

# **16.2** ADVERSE EVENTS

Adverse Events (AEs) will be coded using MedDRA version 16.0. For an individual patient, only adverse events commencing after first dose of IMP and no later than last dose of IMP+1day will be included in the AE and serious adverse event (SAE) summaries. AEs that began prior to the first dose of IMP or more than one day after the final dose of IMP will not be included in the analysis. Where an AE start date is partially or completely missing, and it is unclear using partial dates as to whether the AE is treatment-emergent, it will be assumed that it is.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005

Effective Date: 01May2012 



### 16.2.1 ADVERSE EVENTS

An overall AE summary presenting the number and percentage of patients within the following categories by treatment sequence group and total will be provided.

- Total number of AEs (each patient might be counted more than once within this item)
- Patients with AEs
- Patients with SAEs
- Patients with AEs with a relationship to IMP as "Possible", "Probable" and "Certain"
- Patients with severe AEs
- Patients with AEs leading to IMP dose change
- Patient with AEs leading to IMP permanently discontinued

In addition, an analysis using McNemar's test to compare the AE incidence during the 4-hour post dosing period between treatments will be presented for the following categories:

- Total number of AEs (note that for this item only the total numbers will be presented, no comparison on McNemar's test will be performed)
- Patients with AEs
- Patients with SAEs
- Patients with AEs with a relationship to IMP as "Possible", "Probable" and "Certain"
- Patients with severe AEs

Effective Date: 01May2012

In addition, following tables will be reported by treatment sequence group:

- AEs, by SOC, PT and severity
- Related AEs, by SOC, PT and severity

The tables above will be repeated for adverse events occur during the 4 hour post dosing period by treatment.

Individual listings on adverse events, related adverse events (see definition in section 16.1.1.2), serious adverse events, adverse events leading to dose change/study discontinuation and death will be reported.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005








#### 16.2.1.1 Severity

Severity is classified as mild/ moderate/ severe. AEs with a missing severity will be counted in a separate missing category. If a patient reports an AE more than once within that SOC/ PT, the AE with the worst case severity will be used in the corresponding severity summaries.

#### 16.2.1.2 Relationship to Study Medication

Relationship, as indicated by the Investigator, is classed as "Unassessable/Unclassified", "Conditional/Unclassified", "Unrelated", "Unlikely", "Possible", "Probable", and "Certain". Adverse events with a relationship of "Possible", "Probable" and "Certain" to IMP will be considered as related to study medication. AEs with a missing relationship to study medication will be counted in a separate missing category. If a patient reports the same AE more than once within that SOC/ PT, the AE with the worst case relationship to study medication will be used in the corresponding relationship summaries.

### 16.2.2 Adverse Events Leading to Dose Change or Discontinuation of Study Medication

If the action taken for an AE is recorded as "IMP permanently discontinued" on AE page of the CRF it will be considered as an AE leading to permanent discontinuation. If the action taken for an AE is recorded as "IMP dose changed" on AE page of the CRF it will be considered as an AE leading to dose change. These will be summarized by SOC and PT by treatment sequence group and also listed.

#### 16.2.3 SERIOUS ADVERSE EVENTS

SAEs are those events recorded as "Serious" on the Adverse Events page of the CRF. A summary of SAEs by SOC, PT and severity, as well as a summary of related SAEs by SOC, PT, and severity will be reported by treatment sequence group. The tables will be repeated for serious adverse events during the 4 hour post doing period. Summaries will also be provided for SAEs leading to dose change as well as study discontinuation. These data will also be listed.

#### 16.2.4 Adverse Events Leading to Death

AEs leading to Death are those events with outcome reported as "Fatal" in the Adverse Events page of the CRF. A summary of AEs leading to death by SOC and PT will be prepared. This information will also be listed.

## **16.3 DEATH**

As only AEs leading to death are recorded for this study, please refer to Section 16.1.4.

Reckitt Benckiser GA1202 Statistical Analysis Plan Document:

Author: Version Number: Final 5.1 Version Date: [25Feb2014]

Template No: CS TP BS016 - Revision 3 Reference: CS WI BS005

 Effective Date: 01May2012





# **16.4 LABORATORY EVALUATIONS**

Clinical assessments on hematology and clinical chemistry are to be measured at Visit 1 and Visit 3 (Early Termination Visit). A list of laboratory assessments to be included in the outputs is provided in appendix 1.

Local laboratories will be used for the assessment of hematology and clinical chemistry data and these data will be converted to the International System (SI) of units by Data Management Team using standard conversion factors. Quantitative laboratory measurements reported as "< X", i.e. below the lower limit of quantification (BLQ), or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

At each visit, summary statistics for the absolute laboratory value and the changes from baseline will be presented by treatment sequence group and overall. The significance of changes from baseline will be assessed using the Wilcoxon Signed-Rank Test within each sequence group and overall.

Each pre-study baseline laboratory value will be categorised as low, normal, or high based on the reference range:

Low: Below the lower limit of the laboratory reference range.

Normal: Within the laboratory reference range (upper and lower limit included).

High: Above the upper limit of the laboratory reference range.

Each post-baseline value will be classified in a similar manner, producing a 3 x 3 table for each treatment sequence group at each post-baseline visit. Scores of "1" will be assigned to low values, "2" to normal values, and "3" to high values. Using these scores, shifts from baseline will also be assigned a score. For example, a laboratory value that shifts from low to high will be assigned a score of 2, whilst a laboratory value that remains at a low value will be assigned a score of 0. Shifts between these categories between baseline and Visit 3 (Early Termination Visit) will be compared using the Wilcoxon Signed-Rank test within each treatment sequence group and overall. Statistical testing will be performed at last visit.

In addition to the high and low quantitative laboratory assignments (as identified by means of the laboratory reference ranges), clinically significant quantitative laboratory assessments will be identified by investigator and the result will be recorded in the CRF. The number and percentage of patients with abnormal or clinically significant results will be tabulated by treatment sequence groups by visit. The results will also be listed.

Women of child-bearing potential will undergo urine pregnancy testing (positive or negative). The results will be listed.

# 16.5 ECG EVALUATIONS

Effective Date: 01May2012

A 12-lead ECG examination will be conducted at baseline. The results will be listed and summarised as per Section 10.

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






# 16.6 VITAL SIGNS

Vital signs will be conducted at baseline and final or early termination visits. The following Vital Signs measurements will be reported:

Systolic and diastolic blood pressure (after sitting for 5 minutes; mmHg)

Heart rate (radial pulse counted for 30 seconds after resting for 5 minutes; beats/minute)

At each visit, summary statistics for the absolute vital sign value and the changes from baseline will be presented by treatment sequence group and overall. The significance of changes (within each sequence separately and overall) from baseline will be assessed at the last visit, using the Wilcoxon Signed-Rank Test.

A complete listing on all patients' vital sign result will be presented.

# 16.7 PHYSICAL EXAMINATION

A physical examination is to be performed at Visit 1 and Visit 3 or early termination visit. The following summaries will be provided for physical examination data:

Incidence of clinically significant abnormalities at screening

Incidence of clinically significant abnormalities at Visit 3 (early termination visit)

A shift table on clinically significant abnormalities between baseline and Visit 3 (Early Termination Vist) will be presented, and P- values from McNemar's test will be reported within each sequence group and overall.

A listing on clinical significant abnormalities will be reported.

# 16.8 REFERENCES

1. Reckitt Benckiser GA1202 Study Protocol Final Version 2.0, Amendment 1, 4Jun2013.

## 17 LIST OF TABLES

Effective Date: 01May2012

- 14.1.1 Patient Disposition and Withdrawals All Patients
- 14.1.2 Protocol Deviations/Violations Full Analysis Set
- 14.1.3 Summary of Patiens Excluded from Analysis Populations Full Analysis Set
- 14.1.4 Demographic and Baseline Characteristics Full Analysis Set
- 14.1.5 Smoking habits and Alcohol/Drug Use Full Analysis Set
- 14.1.6 GERD Status at Baseline Full Analysis Set
- 14.1.7 12-Lead ECG Examination Full Analysis Set
- 14.1.8 Endoscopy Examination Full Analysis Set
- 14.1.9.1 Medical History Full Analysis Set
- 14.1.9.2 Concomitant Illnesses Full Analysis Set

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






- 14.1.10.1 Prior Medications and Therapies Full Analysis Set
- 14.1.10.2 Concomitant Medications and Therapies Full Analysis Set
- 14.1.11 NIMP Accountability Safety Population
- 14.1.12 4-Hour Monitoring Procedure Intent-to-treat Population
- 14.2.1.1 Summary of 4-hour pH Monitoring Results based on Adjusted 4-hour Data Intent-to-treat Population
- 14.2.1.2 Summary of 4-hour pH Monitoring Results based on Adjusted 4-hour Data by Center Intent-to-treat Population
- 14.2.2.1 Analysis of Treatment Difference during the 4-hour Post Dosing Period based on Adjusted 4-hour Data -Intent-to-treat Population
- 14.2.2.2 Analysis of Treatment Difference during the 4-hour Post Dosing Period Per protocol Population
- 14.2.2.3 Analysis of Treatment Difference during the 4-hour Post Dosing Period based on Log Transformed Adjusted 4-hour Data - Intent-to-treat Population
- 14.2.3.1 Analysis of Visit and Sequence Difference during the 4-hour Post Dosing Period Intent-to-treat
- 14.2.3.2 Analysis of Visit and Sequence Difference during the 4-hour Post Dosing Period Per Protocol Population
- 14.3.1.1 Summary of All Adverse Events Safety Population
- 14.3.1.2 Comparison of Adverse Events during the 4-hour Post Dosing Period Safety Population
- 14.3.2.1 Overall Adverse Events by System Organ Class, Preferred Term and Intensity Safety Population
- 14.3.2.2 Overall Related Adverse Events by System Organ Class, Preferred Term and Intensity Safety Population
- 14.3.2.3 Overall Serious Adverse Events by System Organ Class, Preferred Term and Intensity Safety Population
- 14.3.2.4 Overall Related Serious Adverse Events by System Organ Class, Preferred Term and Intensity Safety **Population**
- 14.3.2.5 Adverse Events during the 4-hour Post Dosing Period by System Organ Class, Preferred Term and Intensity - Safety Population
- 14.3.2.6 Related Adverse Events during the 4-hour Post Dosing Period by System Organ Class, Preferred Term and Intensity – Safety Population
- 14.3.2.7 Serious Adverse Events during the 4-hour Post Dosing Period by System Organ Class, Preferred Term and Intensity – Safety Population
- 14.3.2.8 Related Serious Adverse Events during the 4-hour Post Dosing Period by System Organ Class, Preferred Term and Intensity – Safety Population
- 14.3.2.9 Adverse Events Leading to Dose Change by System Organ Class and Preferred Term Safety Population
- 14.3.2.10 Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term Safety Population
- 14.3.2.11 Adverse Events Leading to Death Safety Population
- 14.3.2.12 Serious Adverse Events Leading to Dose Change by System Organ Class and Preferred Term Safety Population
- 14.3.2.13 Serious Adverse Events Leading to Study Discontinuation Safety Population
- 14.3.3.1 Hematology: Observed Values Safety Population
- 14.3.3.2 Hematology: Change from Baseline at Visit 3 Safety Population
- 14.3.3.3 Clinical Chemistry: Observed Values Safety Population
- 14.3.3.4 Clinical Chemistry: Change from Baseline at Visit 3 Safety Population

Reckitt Benckiser GA1202 Statistical Analysis Plan Document:

Author: Version Number: Final 5.1 Version Date: [25Feb2014]

Template No: CS TP BS016 - Revision 3 Reference: CS WI BS005


Effective Date: 01May2012





- 14.3.3.5 Abnormal Results in Hematology Safety Population
- 14.3.3.6 Abnormal Results in Clinical Chemistry Safety Population
- 14.3.3.7 Clinically Significant Results in Hematology Safety Population
- 14.3.3.8 Clinically Significant Results in Clinical Chemistry Safety Population
- 14.3.3.9 Shift Table for Hematology Safety Population
- 14.3.3.10 Shift Table for Clinical Chemistry Safety Population
- 14.3.4.1 Vital Signs: Observed Values Safety Population
- 14.3.4.2 Vital Signs: Change from Baseline at Visit 3 Safety Population
- 14.3.5.1 Summary of Physical Examination Results Safety Population
- 14.3.5.2 Shift Table for Physical Examination Safety Population

# 18 LIST OF LISTINGS

- 16.2.1.1 Patient Completion Information All Patients
- 16.2.1.2 Inclusion/Exclusion Criteria Eligibility All Patients
- 16.2.1.3 Population Classification Full Analysis Set
- 16.2.2. Major Protocol Deviations/Violations Full Analysis Set
- 16.2.3.1 Demographic Data Full Analysis Set
- 16.2.3.2 Medical History Full Analysis Set
- 16.2.3.3 Concomitant Illnesses Full Analysis Set
- 16.2.3.4 Smoking Habits and Alcohol/Drug Use Full Analysis Set
- 16.2.3.5 GERD Status at Baseline Full Analysis Set
- 16.2.3.6.1 Prior Medication and Therapies Full Analysis Set
- 16.2.3.6.2 Concomitant Medications and Therapies Full Analysis Set
- 16.2.3.7 Pregnancy Test Results Full Analysis Set
- 16.2.3.8 12-lead ECG at Baseline Full Analysis Set
- 16.2.3.9 Endoscopy Examination Full Analysis Set
- 16.2.3.10 NIMP Accountability Safety Population
- 16.2.4.1 4-hour pH Monitoring Procedure Full Analysis Set
- 16.2.4.2 4-hour pH Monitoring Results Full Analysis Set
- 16.2.5.1 Adverse Events Safety Population
- 16.2.5.2 Related Adverse Events Safety Population
- 16.2.5.3 Serious Adverse Events Safety Population
- 16.2.5.4 Severe Adverse Events Safety Population
- 16.2.5.5 Adverse Events Leading to Dose Change Safety Population
- 16.2.5.6 Adverse Events Leading to Study Discontinuation Safety Population
- 16.2.5.7 Serious Adverse Events Leading to Dose Change Safety Population
- 16.2.5.8 Serious Adverse Events Leading to Study Discontinuation Safety Population
- 16.2.5.9 Death Safety Population

Effective Date: 01May2012

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






- 16.2.6.1 Hematology Results Safety Population
- 16.2.6.2 Clinically Significant Hematology Results Safety Population
- 16.2.6.3 Clinical Chemistry Results Safety Population
- 16.2.6.4 Clinically Significant Chemistry Results Safety Population
- 16.2.7.1 Vital Signs Safety Population
- 16.2.7.2 Physical Examinations Safety Population

# **APPENDIX 1 LIST OF LABORATORY ASSESSMENTS**

# Site 01

Effective Date: 01May2012

Reckitt Benckiser GA1202 Statistical Analysis Plan Document:

Author: Version Number: Final 5.1 Version Date: [25Feb2014]

Template No: CS\_TP\_BS016 - Revision 3 Reference: CS\_WI\_BS005






| Assessment | Normal Range | SI Unit |
|---|---|---|
| Haematology | | |
| Haemoglobin | 113-151 for female, 131-172 for male | g/L |
| Red blood cells | 3.68-5.13 for female, 4.09-5.74 for male | 10^12/L |
| Mean cell haemoglobin concentration | 322-362 for female, 320-355 for male | g/L |
| White blood cells | 3.69-9.16 for female, 3.97-9.15 for male | 10^9/L |
| Platelet count | 101-320 for female, 85-303 for male | 10^9/L |
| Clinical chemistry | | |
| Sodium | 130-147 | mmol/L |
| Potassium | 3.5-5.1 | mmol/L |
| Calcium | 2-2.75 | mmol/L |
| Urea | 2.5-7.1 | mmol/L |
| Creatinine | 53-97 for female, 62-115 for male | μmol/L |
| Uric Acid | 160-430 | μmol/L |
| Glucose | 3.9-6.1 | mmol/L |
| Inorganic phosphorous | 0.8-1.6 | mmol/L |
| Alanine transaminase | 10-64 | U/L |
| Aspartate transaminase | 8-40 | U/L |

# Site 02

Effective Date: 01May2012

| Assessment | Normal Range | SI Unit |
|------------|--------------|---------|

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005






| Haematology | | |
|-------------------------------------|-----------|---------|
| Haemoglobin | 110-170 | g/L |
| Red blood cells | 4.09-5.74 | 10^12/L |
| Mean cell haemoglobin concentration | 320-355 | g/L |
| White blood cells | 3.97-9.15 | 10^9/L |
| Platelet count | 85-303 | 10^9/L |
| Clinical chemistry | | |
| Sodium | 135-145 | mmol/L |
| Potassium | 3.5-5.5 | mmol/L |
| Calcium | 2-2.5 | mmol/L |
| Urea | 1.7-8.3 | mmol/L |
| Creatinine | 40-110 | μmol/L |
| Uric Acid | 119-428 | μmol/L |
| Glucose | 3.6-6.1 | mmol/L |
| Inorganic phosphorous | 1-1.6 | mmol/L |
| Alanine transaminase | 0-75 | U/L |
| Aspartate transaminase | 0-40 | U/L |
| | 1 | 1 |

# <u>Site 03</u>

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005

Effective Date: 01May2012





| Assessment | Normal Range | SI Unit |
|---|---|---|
| Haematology | | |
| Haemoglobin | 110-150 for female, 120-160 for male | g/L |
| Red blood cells | 3.5-5 for female, 4-5.5 for male | 10^12/L |
| Mean cell haemoglobin concentration | 310-350 | g/L |
| White blood cells | 4-10 | 10^9/L |
| Platelet count | 100-300 | 10^9/L |
| Clinical chemistry | 1 | |
| Sodium | 135-148 | mmol/L |
| Potassium | 3.5-5.5 | mmol/L |
| Calcium | 2.15-2.62 | mmol/L |
| Urea | 2.5-6.5 | mmol/L |
| Creatinine | 50-110 | μmol/L |
| Uric Acid | 150-420 | μmol/L |
| Glucose | 3.6-6.1 | mmol/L |
| Inorganic phosphorous | 0.82-1.62 | mmol/L |
| Alanine transaminase | 0-64 | U/L |
| Aspartate transaminase | 0-64 | U/L |

Document: Reckitt Benckiser GA1202 Statistical Analysis Plan

Effective Date: 01May2012


Template No: CS\_TP\_BS016 – Revision 3 Reference: CS\_WI\_BS005


| Page 1 | of | 1 |
|--------|----|---|
|--------|----|---|

| Changes to Pla | anned Statistical Analyses I | Form | Page 1 of 1 |
|---|---|---|---|
| Customer: | RB Healthcare | | |
| Protocol No.: | GA1202 | THE PARTY OF THE P | |
| Project Code: | QVA96908 | | |
| Date: | 19/MAR/2014 | | |
| The timing of th | e change(s) was: | | |
| | | for an open-label study) but befo | re completion of the |
| | Statistical Report/Clinical St | | |
| ☐ Afte | r completion of the final Stati | stical Report/Clinical Study Repo | rt |
| Describe the ch | ange(s) required: | | |
| The term "Full A | analysis Set" is to be renamed | the "All Patient Population" | |
| | | hange(s) and who was involved: | |
| The RB Statistic<br>submitted RB str | al Manager () was idy stating that RB had used t | made aware of a comment made<br>he term Full Analysis Set (FAS) i | by the SFDA on a previous nappropriately. |
| Biological Produ<br>examinees in the<br>in GA1202 repressudy is to be rer<br>headed 'All pati-<br>new definition. | acts" the FAS should be represe<br>minimal and reasonable appresent all randomised patients. a<br>med the All Patient Populatients, this heading will now be | Biostatistics for the Clinical Trial<br>tented as follows: "The data set is<br>each from all the randomized exa<br>Therefore RB request that the Fullon (APP). As listings currently in<br>the headed 'All Screened Patients' to | obtained after excluding the minees". However the FAS I Analysis Set (FAS) in this cluding screen failures are prevent confusion with the |
| | 202 SAP the FAS according to<br>change is necessary for this p | o the guidance is represented by the opulation. | ie Intent to Treat (ITT) |
| The group(s) re | sponsible for the change(s) s | and implications for the study: | |
| The RB Statistic<br>Statisticians are<br>explanation in th | al Manager () is re-<br>responsible for updating the T<br>e Statistical and Clinical Repo | sponsible for requesting this chan<br>FLs and ensuring appropriate doc | umentation and |
| analyses | | W. 20 T. Sec. 19 12 | S.V-85111-111 |
| Form completed<br>Title | <u>by</u> :<br>Name | Signature | Date |
| Mgr, Biostatistic | | Signature | Date |
| Form approved b | V: | | |
| Title | Name | Signature | Date |
| Dir, Biostatistics | | | |
| Form approved b | y Customer Representative (it | applicable): | |

Form No: CS\_FM\_BS006 - Revision 4 Effective Date: 01Feb2010

Name

Statistical Manager

Title

Reference: CS\_WI\_BS005

Date

Copyright © 2010 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

Signature

Changes to Planned Statistical Analyses Form

| Customer: | RB Healthcare | | |
|---|---|---|---|
| Protocol No.: | GA1202 | - (1-70) | |
| Project Code: | QVA96908 | STORE | |
| Date: | 08/MAY/2014 | 18414- | |
| Describe the ch 1. Additional at treatment are a 2. Figure of the Describe the pr Requested by RI | Statistical Report/Clinical Statistical Report/Clinical Statistic completion of the final Statistics ange(s) required: nalyses in which erosive/not added to the primary analyse primary endpoint (ITT popocess used to decide on the cost Statistical Manager ( | stical Report/Clinical Study Repor | nteraction with of DADA v placebo. |
| The RB Statistic<br>Statisticians are | al Manager ( is re | and implications for the study:<br>esponsible for requesting this chang<br>requested output and ensuring appi<br>Reports. | ge and Quintile<br>ropriate documentation |
| Form completed | by:<br>Name | Signature | Date |
| Mgr, Biostatistic | | Signature | Date |
| D. 0.885 | | | |
| | The second secon | | |
| | <u></u> | Signature | Data |
| Form approved b | oy:<br>Name | Signature | Date |
| Title | oy:<br>Name | Signature | Date |
| Title<br>Dir, Biostatistics | oy:<br>Name | | Date |
| Title<br>Dir, Biostatistics | oy:<br>Name | | Date Date |

Form No: CS\_FM\_BS006 - Revision 4 Effective Date: 01Feb2010 Reference: CS\_WI\_BS005

Copyright © 2010 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.

| ALC: NO | | | |
|---------|--------|--------|---|
| 2 3 | OIL | 10.170 | - |
| 5 2 | ( )1 1 | INTI | |
| No. | ~~~ | | |

Changes to Planned Statistical Analyses Form

| Customer: | RB Healthcare |
|---|---|
| Protocol No.: | GA1202 |
| Project Code: | QVA96908 |
| Date: | 17/JUL/2014 |
| The timing of the | change(s) was: |
| | r unblinding (or database lock for an open-label study) but before completion of the |
| final Statistical Report/Clinical Study Report | |
| ☐ Afte | r completion of the final Statistical Report/Clinical Study Report |
| Describe the ch | ange(s) required: |
| | g on minor protocol deviation is to be added. |
| Troditional Hoting | , on miles protocol deviation is to be added. |
| Describe the pro | ocess used to decide on the change(s) and who was involved: |
| During the prepa | ration of the Clinical Study Report, the Quintiles Medical Writer ( |
| | e 14.1.2 includes an analysis of the minor protocol deviation, yet the listing referred to |
| (Listing 16.2.2) c | only covers the major deviation. |
| According to the | ICH GCP guidance, it was interpreted that only major deviation need to be reported hence |
| | col deviation listing was included in the SAP. However, to solve the anomaly in the CSR, |
| RB Clinical Man | |
| listing added to d | lisplay the minor deviation. |
| | No. of the second secon |
| | 2.2 will become 16.2.2.1, and a new listing 16.2.2.2 will present all minor protocol |
| deviation. Table | 14.1.2 will reference both listings. |
| The group(s) res | sponsible for the change(s) and implications for the study: |
| The RB Clinical | |
| requesting this cl | nange and Quintile Statisticians are responsible for providing the additional listing and |
| ensuring appropr | iate documentation and explanation in the Statistical and Clinical Reports. |
| Form completed Title | by: |
| AD, Biostatistics | |
| AD, Diostatistics | |
| Form approved b | |
| Title | Name Signature Date |
| Dir, Biostatistics | |
| Form approved b | y Customer Representative (if applicable): |
| Title | Name Circulate Circulate P |
| Statistical Manag | er |

Page 1 of 1

Form No: CS\_FM\_BS006 - Revision 4

Effective Date: 01Feb2010

Reference: CS\_WI\_BS005

Copyright © 2010 Quintiles Transnational Corp. All rights reserved.

The contents of this document are confidential and proprietary to Quintiles Transnational Corp. Unauthorized use, disclosure or reproduction is strictly prohibited.